CLINICAL TRIAL: NCT02375152
Title: Safety and Effectiveness of Capsulotomy in Refractory Obsessive-Compulsive Disorder
Brief Title: Safety and Effectiveness of Capsulotomy in Refractory OCD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Bomin Sun, Director of the Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-14
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: neurosurgery; capsulotomy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical Intervention (Experimental)
  Interventions: Procedure: Anterior Capsulotomy

INTERVENTIONS:
Procedure: Anterior Capsulotomy

SUMMARY:
Obsessive-compulsive disorder (OCD) is a severely disabling psychiatric disorder with a worldwide lifetime prevalence of 2-3% (Islam et al., 2015).Despite the efficacy of pharmacological and behavioural treatment methods for most OCD patients, roughly one third do not demonstrate significant symptom improvement, even after aggressive treatment (Foa et al, 2007). The effectiveness of neurosurgical treatment methods (including ablative surgery) for those with severely disabling treatment resistant OCD is substantiated by clinical research (Greenberg, Rauch & Haber, 2010). The brain target of this procedure is usually the area between the anterior and middle third of the anterior limb of the internal capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Obsessive compulsive disorder as the primary psychiatric diagnosis (according to DSM IV-criteria).
2. Severity: Score higher than 25 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS).
3. Course of illness had to have been present for at least five years in a chronic or progressive form despite any treatment trials (refractory).
4. Refractory: a lack of response to drug therapy after adequate administration (defined as more than 12 weeks at the maximum tolerated dose) of at least three serotonin-reuptake inhibitors, and clomipramine. Adequate psychotherapy, defined as continuously treatment for more than six months with a certified therapist .

Exclusion Criteria:

1. Schizophrenic disorder; bipolar disorder; substance abuse or dependence (except for dependence on nicotine), as assessed with the use of the Mini-International Neuropsychiatric Interview (MINI 6.0.0);
2. Cluster A or B personality disorder according to DSM-IV criteria, as assessed with the use of the Structured Clinical Interview II.
3. A current severe major depressive episode, determined according to DSM-IV criteria (as assessed with the use of the MINI 6.0.0) and defined by HAMD-17 score of more than 20 and a risk of suicide.
4. Abnormal cognitive status (measured by MoCA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Y-BOCS Score | Baseline (preoperative), 3 months, 6 months

SECONDARY OUTCOMES:
Change in Clinical Global Impressions Scale Score | Baseline (preoperative), 3 months, 6 months
Change in Hamilton Anxiety Scale, Hamilton Depression Scale-17 Score | Baseline (preoperative), 3 months, 6 months
Change in Temperament and Character Inventory revised version (TCI-R) Score | Baseline (preoperative), 3 months, 6 months
Change in functional magnetic resonance imaging (fMRI) images | Baseline (preoperative), 3 months, 6 months
Change in Psychophysical tasks（ Iowa Gambling Task , Model Task, Working memory task ） | Baseline (preoperative), 3 months, 6 months
WHO disability assessment 2.0 (self, 12 terms) | Baseline (preoperative), 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Greenberg BD, Gabriels LA, Malone DA Jr, Rezai AR, Friehs GM, Okun MS, Shapira NA, Foote KD, Cosyns PR, Kubu CS, Malloy PF, Salloway SP, Giftakis JE, Rise MT, Machado AG, Baker KB, Stypulkowski PH, Goodman WK, Rasmussen SA, Nuttin BJ. Deep brain stimulation of the ventral internal capsule/ventral striatum for obsessive-compulsive disorder: worldwide experience. Mol Psychiatry. 2010 Jan;15(1):64-79. doi: 10.1038/mp.2008.55. Epub 2008 May 20. PMID 18490925
- [Background] Foa EB, Liebowitz MR, Kozak MJ, Davies S, Campeas R, Franklin ME, Huppert JD, Kjernisted K, Rowan V, Schmidt AB, Simpson HB, Tu X. Randomized, placebo-controlled trial of exposure and ritual prevention, clomipramine, and their combination in the treatment of obsessive-compulsive disorder. Am J Psychiatry. 2005 Jan;162(1):151-61. doi: 10.1176/appi.ajp.162.1.151. PMID 15625214
- [Background] Pepper J, Hariz M, Zrinzo L. Deep brain stimulation versus anterior capsulotomy for obsessive-compulsive disorder: a review of the literature. J Neurosurg. 2015 May;122(5):1028-37. doi: 10.3171/2014.11.JNS132618. Epub 2015 Jan 30. PMID 25635480